CLINICAL TRIAL: NCT01513759
Title: A Prospective, Single-Arm, Multi-Center Trial of EkoSonic® Endovascular System and Activase for Treatment of Acute Pulmonary Embolism (PE)
Brief Title: Submassive and Massive Pulmonary Embolism Treatment With Ultrasound Accelerated Thrombolysis Therapy
Acronym: SEATTLE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKOS 09
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Embolism; Acute Pulmonary Embolism; Sub-massive Pulmonary Embolism; Massive Pulmonary Embolism; Pulmonary Thromboembolism
Keywords: Fibrinolysis; catheter directed fibrinolysis; ultrasound accelerated fibrinolysis; recombinant t-PA; Activase
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EkoSonic® Endovascular System (Experimental): Participants will receive a total of 24 milligrams (mg) of recombinant t-PA infusion, at an infusion rate of 1 milligrams/hour (mg/hr) per device (2 mg/hour for bilateral PE) delivered through the EkoSonic® Endovascular System. This regimen allows for a recombinant t-PA infusion time of 24 hours for one catheter and 12 hours for two catheters, respectively.
  Interventions: Drug: recombinant tissue plasminogen activator; Device: EKOS EkoSonic Endovascular System

INTERVENTIONS:
Drug: recombinant tissue plasminogen activator — Participants will receive 24 mg of r-tPA delivered via the EkoSonic Endovascular Device.
  Other Names: r-tPA; t-PA; Alteplase
Device: EKOS EkoSonic Endovascular System — 24 mg of r-tPA will be delivered through the EkoSonic Endovascular System.
  Other Names: EkoSonic Endovascular Device; EkoSonic

SUMMARY:
The purpose of this study is to determine if the EKOS EkoSonic® Endovascular Device when used in conjunction with recombinant tissue plasminogen activator (t-PA) as a treatment for acute PE will decrease the ratio of right ventricle (RV) to left ventricle (LV) diameter within 48 =/- 6 hours in participants with massive or submassive PE.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography (CT) evidence of proximal PE (filling defect in at least one main or segmental pulmonary artery)
* PE symptom duration less than or equal to (<=)14 days
* Informed consent can be obtained from participant or Legally Authorized Representative (LAR)
* Massive PE (syncope, systemic arterial hypotension, cardiogenic shock, or resuscitated cardiac arrest) or
* Submassive PE (RV diameter-to-LV diameter greater than or equal to [>=] 0.9 on contrast-enhanced chest CT)

Exclusion Criteria:

* Stroke or transient ischemic attack (TIA), head trauma, or other active intracranial or intraspinal disease within one year
* Recent (within one month) or active bleeding from a major organ
* Hematocrit less than (<) 30 percent (%)
* Platelets < 100 thousand/microliter (mcL)
* International Normalized Ratio (INR) greater than (>) 3
* Activated partial thromboplastin time (aPTT) >50 seconds on no anticoagulants
* Major surgery within seven days of screening for study enrollment
* Serum creatinine >2 milligrams/deciliter (mg/dL)
* Clinician deems high-risk for catastrophic bleeding
* History of heparin-induced thrombocytopenia (HIT)
* Pregnancy
* Catheter-based pharmacomechanical treatment for pulmonary embolism within 3 days of study enrollment
* Systolic blood pressure less than 80 mm Hg despite vasopressor or inotropic support
* Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR)
* Evidence of irreversible neurological compromise
* Life expectancy <30 days
* Use of thrombolytics or glycoprotein IIb/IIIa antagonists within 3 days prior to inclusion in the study
* Previous enrollment in the SEATTLE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2013-02-17 (Actual); Study Completion 2013-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Bhalla, MD, Principal Investigator — Baptist Health; William Kuo, MD, Principal Investigator — Stanford Hospital and Clinics; Stephen K Liu, MD, Principal Investigator — Memorial Medical Center - Modesto; Immad Sidiq, MD, Principal Investigator — Hartford Hospital; Samuel Z Goldhaber, MD, Study Chair — Brigham and Women's; Mark J Garcia, MD, Principal Investigator — Christiana Hospital; Rohit Bhatheja, MD, Principal Investigator — AdventHealth; Robert Kennedy, MD, Principal Investigator — Holmes Regional Medical Center; Fakhir Elmasri, MD, Principal Investigator — Lakeland Regional Medical Center; Barry S Weinstock, MD, Principal Investigator — Orlando Regional Medical Center; Juan Ayerdi, MD, Principal Investigator — Medical Center of Central Georgia; Nilesh Goswami, MD, Principal Investigator — Prairie Heart Institute - St.John's Hospital; Kannan Natarajan, MD, Principal Investigator — St Vincent's Hospital; Tod C Engelhardt, MD, Principal Investigator — East Jefferson General Hospital; Mark Kumar, MD, Principal Investigator — Overlook Medical Center; John Rundback, MD, Principal Investigator — Holy Name Hospital; Jacob Cynamon, MD, Principal Investigator — Montefiore Medical Center; Peter Soukas, MD, Principal Investigator — The Miriam Hospital; Mohammad L Raja, MD, Principal Investigator — Providence Memorial Hospital - Sierra Vista Hospital; Keith M Sterling, MD, Principal Investigator — Inova Alexandria; John Gurley, MD, Principal Investigator — University of Kentucky; Noah Jones, MD, Principal Investigator — Mt. Carmel East
Locations (22):
- United States (22):
  - Baptist Health, Montgomery, Alabama
  - Memorial Medical Center, Modesto, California
  - Stanford University Medical Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Prairie Heart Institute, Springfield, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - University of Kentucky, Gill Heart Institute, Lexington, Kentucky
  - East Jefferson General Hospital, New Orleans, Louisiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Overlook Medical Center, Morristown, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Mt. Carmel East, Columbus, Ohio
  - The Miriam Hospital, Providence, Rhode Island
  - Providence Memorial and Sierra Medical Center, El Paso, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia

REFERENCES:
- [Derived] Sadiq I, Goldhaber SZ, Liu PY, Piazza G; Submassive and Massive Pulmonary Embolism Treatment with Ultrasound AcceleraTed ThromboLysis ThErapy (SEATTLE II) Investigators. Risk factors for major bleeding in the SEATTLE II trial. Vasc Med. 2017 Feb;22(1):44-50. doi: 10.1177/1358863X16676355. Epub 2017 Jan 31. PMID 27913777
- [Derived] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743

RESULTS

PARTICIPANT FLOW:
Groups:
- EkoSonic® Endovascular System: Participants received a total of 24 milligrams (mg) of recombinant tissue plasminogen activator (r-tPA) infusion, at an infusion rate of 1 milligrams/hour (mg/hr) per device (2 mg/hour for bilateral pulmonary embolism [PE]) delivered through the EkoSonic® Endovascular System. This regimen allowed for a r-tPA infusion time of 24 hours for one catheter and 12 hours for two catheters, respectively.
Period: Overall Study
Arm/Group | EkoSonic® Endovascular System
Started | 150
At Least One Device Successfully Placed | 149
Completed | 145
Not Completed | 5
Not completed — Protocol Violation | 4
Not completed — Death during catheter placement | 1

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set included all participants who started the ultrasound accelerated thrombolysis therapy.
Groups:
- EkoSonic® Endovascular System: Participants received a total of 24 mg of r-tPA infusion at an infusion rate of 1 mg/hr per device (2 mg/hour for bilateral PE) delivered through the EkoSonic® Endovascular System. This regimen allowed for a r-tPA infusion time of 24 hours for one catheter and 12 hours for two catheters, respectively.
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, Not of Hispanic Origin | 119
  African American, Not of Hispanic Origin | 22
  Hispanic or Latino | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Right Ventricle (RV) Diameter-to-Left Ventricle (LV) Diameter Ratio Within 48 +/- 6 Hours of Initiation of Therapy
Description: Change from baseline in RV diameter/LV diameter ratio was determined by contrast-enhanced chest computed tomography (CT) within 48 +/- 6 hours after initiating ultrasound-accelerated catheter-directed fibrinolysis.
Time Frame: Baseline, within 48 +/- 6 hours of initiation of therapy
Population: Efficacy analysis set included all participants who started the ultrasound accelerated thrombolysis therapy. Here, 'Overall number of participants analyzed' signifies participants with available data at both baseline and post-baseline. 'Number analyzed' signifies participants with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- EkoSonic® Endovascular System: Participants received a total of 24 mg of r-tPA infusion, at an infusion rate of 1 mg/hr per device (2 mg/hour for bilateral PE) delivered through the EkoSonic® Endovascular System. This regimen allowed for a r-tPA infusion time of 24 hours for one catheter and 12 hours for two catheters, respectively.
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 150
ratio
  Baseline: number analyzed (Participants) | 123
  Baseline | 1.55 (0.39)
  Change within 48 +/- 6 hours: number analyzed (Participants) | 115
  Change within 48 +/- 6 hours | -0.42 (0.36)

2. Primary Outcome: Number of Participants With Major Bleeding
Description: Bleeding adverse events were graded (severe or life-threatening, moderate or mild bleeding) according to the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) classification. The participant incidence of major bleeding events was defined as GUSTO moderate and severe events occurring within 72 hours after starting the ultrasound-accelerated catheter-directed fibrinolysis procedure. Mild: Does not meet criteria for moderate or severe; Moderate: Requires transfusion - No hemodynamic compromise; and Severe: Bleeding causes hemodynamic compromise and required intervention or intracranial hemorrhage. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From start of study drug infusion up to 72 hours
Population: Safety analysis set included all participants who started the EkoSonic device placement procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 150
Participants | 14

3. Secondary Outcome: Change From Baseline in Pulmonary Artery Systolic Pressure at 48 Hours After Start of Therapy
Description: Change in pulmonary artery systolic pressure was assessed by baseline right-heart catheterization compared with right-heart catheterization at the conclusion of ultrasound-accelerated catheter-directed fibrinolysis and estimated by post-procedure transthoracic echocardiography within 48 hours after initiating the procedure.
Time Frame: Baseline, Hour 48 after initiation of therapy
Population: Efficacy analysis set included all participants who started the ultrasound accelerated thrombolysis therapy. Here, 'Number analyzed' signifies participants with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 150
millimeters of mercury (mmHg)
  Baseline | 51.4 (16)
  Change at Hour 48: number analyzed (Participants) | 98
  Change at Hour 48 | -14.4 (15.4)

4. Secondary Outcome: Percentage of Participants With Symptomatic Recurrent Pulmonary Embolism (PE)
Description: Percentage of participants with symptomatic recurrent PE up to 30 days following the conclusion of the ultrasound-accelerated catheter-directed fibrinolysis procedure, were reported with a Wilson score 95% confidence interval. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 30
Population: Efficacy analysis set included all participants who started the ultrasound accelerated thrombolysis therapy. One participant was excluded from this analysis due to lost to follow-up after discharge.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 149
percentage of participants | 0 [0 to 2.5]

5. Secondary Outcome: Number of Participants Who Died Due to Any Cause
Description: Number of participants who died due to any cause for up to 30 days following the conclusion of the ultrasound-accelerated catheter-directed fibrinolysis procedure, were reported.
Time Frame: Baseline up to Day 30
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 149
Participants | 4

6. Secondary Outcome: Number of Devices That Could Not be Successfully Used for Infusion
Description: Technical complications associated with the use of the EkoSonic device was recorded during catheter placement in the pulmonary artery and during the infusion procedure.
Time Frame: Baseline up to Day 30
Population: Safety analysis set included all participants who started the EkoSonic device placement procedure.
Measure: Count of Units; unit: devices
Units Other Than Participants: devices
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 150
Number analyzed (devices) | 285
devices | 7

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30
Description: Safety analysis set included all participants who started the EkoSonic device placement procedure.
Arm/Group | EkoSonic® Endovascular System
Serious Adverse Events (participants affected / at risk) | 28/150
Other Adverse Events (participants affected / at risk) | 59/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EkoSonic® Endovascular System (N=150)
Anemia (Blood and lymphatic system disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Chest Pain (General disorders) | 1
Sepsis (Infections and infestations) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 3
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Electroencephalogram abnormal (Investigations) | 1
Renal failure acute (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Haematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EkoSonic® Endovascular System (N=150)
Anemia (Blood and lymphatic system disorders) | 6
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 4
Chest pain (Cardiac disorders) | 1
Pyrexia (Cardiac disorders) | 2
Cellulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 5
Arterial injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Convulsion (Nervous system disorders) | 1
Haematoma (Vascular disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Haematuria (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Mental status changes (Psychiatric disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Renal failure chronic (Renal and urinary disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days